CLINICAL TRIAL: NCT03990909
Title: A Pilot Study of Dietary Supplementation With Branched Chain Amino Acids on Sleep
Brief Title: Pilot Study of BCAA on Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miranda M Lim, Principal Investigator, Portland VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIRB 4312
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Sleep Wake Disorders; Brain Injuries, Traumatic | interventions — Amino Acids; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCAAs (Experimental): 60 grams of BCAA (2:1:1 ratio of Leucine:Isoleucine:Valine) consumed in two doses (30 grams each) mixed into 20 oz of water for up to 21 days (42 total drinks).
  Interventions: Dietary Supplement: Branched Chain Amino Acids
- Rice Protein (Placebo Comparator): Rice protein control group: 60 grams of rice protein consumed in two doses (30 grams each) mixed into 20 oz of water for up to 21 days (42 total drinks).
  Interventions: Dietary Supplement: Rice Protein
- Microcrystalline Cellulose (Placebo Comparator): Placebo control group: 60 grams of microcrystalline cellulose, consumed in two doses (30 grams each) mixed into 20 oz of water for up to 21 days (42 total drinks).
  Interventions: Dietary Supplement: Microcrystalline Cellulose

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acids — 60 grams of BCAA (2:1:1 ratio of Leucine:Isoleucine:Valine) consumed in two doses (30 grams each) mixed into 20 oz of water for up to21days (42 total drinks).
  Other Names: BCAAs
  Arms: BCAAs
Dietary Supplement: Rice Protein — 60 grams of rice protein consumed in two doses (30 grams each) mixed into 20 oz of water for up to 21days (42 total drinks).
  Arms: Rice Protein
Dietary Supplement: Microcrystalline Cellulose — 60 grams of microcrystalline cellulose, consumed in two doses (30 grams each) mixed into 20 oz of water for up to 21days (42 total drinks).
  Arms: Microcrystalline Cellulose

SUMMARY:
Individuals will be recruited from the VA Portland Health Care System and the community affiliated with Oregon Health & Science University. Traumatic brain injury status will be assessed as a contributing factor. Subjects will be randomized to one of 3 groups (BCAA or one of 2 placebo conditions) and instructed to consume study product twice daily for 21 days. Self-report questionnaires, wrist actigraphy, pressure pain testing, and cognitive function will be assessed pre and post the experimental period.

DETAILED DESCRIPTION:
The goal of this proposal is to explore the feasibility of, and potential for, dietary supplementation with branched chain amino acids (BCAAs) to effect sleep quality and cognitive function in Veterans. The BCAAs (Leucine, Isoleucine, and Valine) cannot be synthesized endogenously (i.e., they must be obtained through the diet) and are the precursors to >50% of de novo glutamate and GABA synthesis in the brain, which are the primary excitatory and inhibitory neurotransmitters, respectively. Preclinical evidence strongly suggests that dietary BCAA supplementation restores normal sleep-wake patterns and cognitive function following TBI through a restoration in the global cortical excitation:inhibition ratio. BCAA supplementation has been studied extensively in healthy humans and in a variety of disease states, including following TBI, but not yet in Veterans in the chronic phase of recovery from TBI. BCAAs are a commercially available dietary supplement and very well tolerated with minimal side-effects.

Subjects will be randomized in a double-blind fashion through the VA Research Pharmacy to one of three groups: 1) BCAA; 60 g/day in two 30 g doses, 2) rice protein; 60 g/day in two 30 g doses, and 3) placebo; 60 g microcrystalline cellulose in two 30 g doses. BCAA and placebo will be prepared by the VA Research Pharmacy and dispensed in a blinded fashion to Veterans after demonstrating informed consent. Following a ~4-week period of baseline, Veterans will be instructed to consume study product after waking and ~6 hours later, on an empty stomach for a period of up to 21-days. Self-report questionnaires assessing sleep quality, cognitive function, trauma-related symptom severity, and other measures of mental and physical well-being will be administered before and after the experimental period. Wrist actigraphy will be continuously collected over the baseline and the experimental period. Cognitive function will be assessed before and after the experimental period using an established battery of neuropsychological tests (i.e., selected tests from WAIS, D-KEFS, HVLT, COWAT, among others. Pressure pain testing will be conducted before and after the experimental period.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* English Speaking
* Accessible via phone
* Sleep problems

Exclusion Criteria:

* Decisional impairment
* Nickel allergy
* Maple syrup urine disease or family history of disease
* Allergy to sucralose
* Currently taking BCAAs

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | 5 weeks
  Number enrolled per month, proportion who complete the protocol
Rates of adherence and treatment fidelity | 5 weeks
  Proportion of subjects consuming full doses
Assessment process and patient acceptability | 5 weeks
  Proportion of questionnaires properly completed, actiwatches properly worn, and patient acceptance of protocol

SECONDARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline; after 3 weeks of intervention
  Measures self-reported insomnia severity; total score range = 0-28 (higher total score = worse insomnia)

CONTACTS AND LOCATIONS:
Overall Officials: Miranda M Lim, MD, PhD, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Health Care System, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifiable data will be made available to qualified researchers on request to the study PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Information will be sent as soon as is practical and will be available as long as the PI is available.
Access Criteria: Legitimate research agenda, including but not limited to request to double-check presented or published results and novel analyses.

REFERENCES:
- [Derived] Elliott JE, Keil AT, Mithani S, Gill JM, O'Neil ME, Cohen AS, Lim MM. Dietary Supplementation With Branched Chain Amino Acids to Improve Sleep in Veterans With Traumatic Brain Injury: A Randomized Double-Blind Placebo-Controlled Pilot and Feasibility Trial. Front Syst Neurosci. 2022 May 4;16:854874. doi: 10.3389/fnsys.2022.854874. eCollection 2022. PMID 35602971